CLINICAL TRIAL: NCT01434576
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Pharmacodynamics and Safety of HGS1025, a Human Monoclonal Anti-CCR5 Antibody, in Subjects With Ulcerative Colitis
Brief Title: Study to Evaluate the Pharmacodynamics and Safety of HGS1025 in Patients With Ulcerative Colitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew study for business reasons
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGS1025-C1106
Record Dates: First submitted 2011-09-01; First posted 2011-09-15 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HGS1025 2 mg/kg (Experimental)
  Interventions: Biological: HGS1025
- HGS1025 10 mg/kg (Experimental)
  Interventions: Biological: HGS1025
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HGS1025 — 2 mg/kg of HGS1025 administered by IV infusion on Day 0, 14, 28 and 56, and then every 28 days thereafter if patient achieves clinical response
  Arms: HGS1025 2 mg/kg
Biological: HGS1025 — 10 mg/kg of HGS1025 administered by IV infusion on Day 0, 14, 28 and 56, and then every 28 days thereafter if patient achieves clinical response
  Arms: HGS1025 10 mg/kg
Drug: Placebo — Placebo administered by IV infusion on Day 0, 14, 28 and 56. Subjects receiving placebo during the first 8 weeks of treatment will be given the option to receive HGS1025 10 mg/kg in the continuation phase of the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics, safety, and pharmacokinetics of HGS1025 in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Active, moderate to severe ulcerative colitis (UC) confirmed by endoscopy
* Currently on 1 or more of the following UC treatment medications: 5-aminosalicylates (5-ASA), corticosteroids, azathioprine, 6-mercaptopurine (6MP), and/or other immunosuppressive or immunomodulatory agents including cyclosporine, tacrolimus, methotrexate, and mycophenolic acid
* Not pregnant or nursing
* Females of non-childbearing potential or females of childbearing potential must be willing to practice abstinence from intercourse from 2 weeks prior to first dose of study agent and for 8 weeks after the last dose of study agent or use effective contraception for 1 month prior to the 1st dose of study agent and through 8 weeks after the last dose of study agent
* Males must agree to use effective contraception throughout the study and for 8 weeks after the last dose of study agent
* Have the ability to provide informed consent and comply with study procedures

Exclusion Criteria:

* Received any of the following within 60 days of the first dose of study agent: Anti-TNFα therapy; integrin receptor antagonist; intravenous immunoglobulin; high dose prednisone or prednisone equivalent (greater than 60 mg/day); any investigational agent including immunosuppressive/immunomodulatory or non-biologic agents
* Have had a change in corticosteroid, 5-ASA, or other immunosuppressive/immunomodulatory agents within 30 days of Day 0
* History of liver disease
* History of a major organ transplant
* History of prior large bowel resection
* Current unstable or uncontrolled acute or chronic diseases not due to UC
* History of malignant neoplasm within the last 5 years, except for some types of adequately treated cancers of the skin or carcinoma in situ of the uterine cervix
* Current or recent drug or alcohol abuse or dependence
* History of a positive test for HIV or test positive for Hepatitis B (HBsAg) or Hepatitis C
* Have a history of severe drug allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics (serum & tissue biological markers; CCR5 receptor occupancy) | 8 weeks
  Change in CCR5 properties; change in inflammatory markers in blood and colon.
Clinical Response | 8 weeks
  Decrease in Mayo Score and rectal bleeding.

SECONDARY OUTCOMES:
Type, frequency, and severity of adverse events | Through 8 weeks after the last dose of study agent
Clinical response | 4 weeks
  Decrease in Mayo Score and rectal bleeding.
Clinical remission | 4 weeks & 8 weeks
  Decrease in Mayo Score and no rectal bleeding or colon friability.
Mucosal healing | 4 weeks & 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline